CLINICAL TRIAL: NCT00099749
Title: Safety and Efficacy of FTY720 in Adult Patients Who Receive a Kidney Transplant
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CFTY720A2218
Record Dates: First submitted 2004-12-17; First posted 2004-12-20 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Kidney Transplantation
Keywords: Kidney, immunosuppression, transplant, rejection
MeSH Terms: conditions — Rejection, Psychology | interventions — Fingolimod Hydrochloride

INTERVENTIONS:
Drug: FTY 720

SUMMARY:
The efficacy and safety of FTY720 is being evaluated in patients who receive a kidney transplant.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female
* Between 18 to 65 years old

Exclusion Criteria:

* Patients in need of multiple organ transplants

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 255
Dates: Start 2003-11; Primary Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Biopsy-proven acute rejection (BPAR), graft loss, death and study discontinuation, within 6 months post transplantation.

SECONDARY OUTCOMES:
Safety/tolerability based on adverse event reporting.
BPAR, graft loss, death and study discontinuation, within 6 and 12 months post transplantation.
Efficacy parameters between the 3 treatment groups within 6 and 12 months post-transplantation.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Director — Novartis
Locations (5):
- United States (5):
  - Loyola University Medical Center, Maywood, Illinois
  - SIU School of Medicine, Springfield, Illinois
  - St. Barnabas Medical Center, Livingston, New Jersey
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island

REFERENCES:
- [Result] Tedesco-Silva H, Szakaly P, Shoker A, Sommerer C, Yoshimura N, Schena FP, Cremer M, Hmissi A, Mayer H, Lang P; FTY720 2218 Clinical Study Group. FTY720 versus mycophenolate mofetil in de novo renal transplantation: six-month results of a double-blind study. Transplantation. 2007 Oct 15;84(7):885-92. doi: 10.1097/01.tp.0000281385.26500.3b. PMID 17984842